CLINICAL TRIAL: NCT07148102
Title: Diaphragmatic Ultrasound and Thoracic Fluid Content for Prediction of Non-Invasive Ventilation Failure in Neonates
Status: Completed | Type: Observational
Sponsor: Lamiaa Khaled Zidan (Other)
Responsible Party: Sponsor-Investigator, Lamiaa Khaled Zidan, Lecturer of Pediatrics, Tanta University
Organization: Tanta University (Other)
Other Study IDs: DTF, DE, TFC with NIV failure
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Diaphragm Ultrasound; Electrical Cardiometry; Non Invasive Ventilation (NIV); RDS of Prematurity
Keywords: EC; NIV; RDS; TFC; DTF; DE
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CPAP: 30 infants supported by nasal CPAP
  Interventions: Device: Diaphragmatic US; Device: EC
- NIPPV: 30 infants supported by non-invasive positive pressure ventilation
  Interventions: Device: Diaphragmatic US; Device: EC
- NHFOV: 30 infants supported with nasal high-frequency oscillatory ventilation
  Interventions: Device: Diaphragmatic US; Device: EC

INTERVENTIONS:
Device: Diaphragmatic US — Diaphragmatic thickening fraction (DTF) and diaphragmatic excursion (DE) were measured by ultrasound within the first three hours of life and repeated either 24 hours later in successful cases or immediately before intubation in cases who had NIV failure.
Device: EC — TFC was assessed using electrical cardiometry (EC). Measurements were obtained within the first three hours of life and repeated either 24 hours later in successful cases or immediately before intubation in cases who had NIV failure.

SUMMARY:
This research assessed diaphragmatic ultrasound and thoracic fluid content (TFC) as potential early predictive tools for detecting NIV failure in preterm neonates.

DETAILED DESCRIPTION:
Non-invasive ventilatory support (NIV) is considered a gold standard care for preterm infants with respiratory distress syndrome (RDS); however, NIV failure remains a frequent challenge that is often associated with many adverse outcomes

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates of both sexes, with gestational ages ranging from 28 to 34 weeks, diagnosed with RDS and requiring non-invasive ventilation within 30 minutes of birth

Exclusion Criteria:

* Exclusion criteria included intubation in the delivery room, complex congenital heart disease, major congenital anomalies in the lungs or airways, and other causes of respiratory distress unrelated to RDS.

Ages: 30 Minutes to 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates (28-34 weeks GA) with RDS and requiring NIV
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
The predictive value | Two years
  The predictive value of DTF, DE, and TFC for NIV failure in preterm neonates with RDS.

SECONDARY OUTCOMES:
Success Rate | Two years
  Comparing success rates among CPAP, NIPPV, and NHFOV groups,

CONTACTS AND LOCATIONS:
Overall Officials: Heba Saied Elmahdy, Professor, Study Director — Faculty of Medicine, Tanta University, Tanta, Q2x2+cp Tanta 2, Egypt, 31527
Locations (1):
- Faculty of Medicine, Tanta University, Tanta, Tanta, Q2x2+cp Tanta 2, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elgendy EM, Elmahdy HS, Nassar MAE, Zidan LK, Eltomey MA, Elsharkawy HM. Diaphragmatic ultrasound and thoracic fluid content for prediction of non-invasive ventilation failure in neonates: a randomized controlled trial. Eur J Pediatr. 2025 Dec 9;185(1):3. doi: 10.1007/s00431-025-06605-8. PMID 41364345